CLINICAL TRIAL: NCT05467306
Title: Enhancing PrEP Outcomes Among Kenyan Adolescent Girls and Young Women With a Novel Pharmacy-based PrEP Delivery Platform
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jillian Pintye, Assistant Professor: Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00013956; R01HD108041 (NIH)
Record Dates: First submitted 2022-07-13; First posted 2022-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-06

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nurse-Navigator Enhanced PrEP Support (Experimental): Pharmacies randomized to the nurse-navigator model will receive tailored support counseling, in addition to receipt of standard PrEP services. Support counseling by nurse-navigators will provide educational messaging tailored to AGYW and actionable advice targeting PrEP persistence and adherence and/or FP topics, and will address participants' questions related to the content. Counseling will include adherence encouragement (IMB domain: motivation), PrEP efficacy and safety (IMB domain: information), self-efficacy for prevention of HIV, support for potential PrEP side effects, behavioral skills (tips for remembering PrEP medications, IMB domain: behavioral skills) and strategies for remembering PrEP refill schedules. During enrollment, the nurse-navigator will explain that support counseling is voluntary and that the nurse will also be available at the pharmacy to address concerns or questions whenever they arise outside of scheduled visits.
  Interventions: Behavioral: Nurse-Navigator Enhanced PrEP Support
- Standard PrEP services (No Intervention): Standard PrEP services

INTERVENTIONS:
Behavioral: Nurse-Navigator Enhanced PrEP Support — Pharmacies randomized to the nurse-navigator model will receive tailored support counseling, in addition to receipt of standard PrEP services. Support counseling by nurse-navigators will provide educational messaging tailored to AGYW and actionable advice targeting PrEP persistence and adherence and/or FP topics, and will address participants' questions related to the content. Counseling will include adherence encouragement (IMB domain: motivation), PrEP efficacy and safety (IMB domain: information), self-efficacy for prevention of HIV, support for potential PrEP side effects, behavioral skills (tips for remembering PrEP medications, IMB domain: behavioral skills) and strategies for remembering PrEP refill schedules. During enrollment, the nurse-navigator will explain that support counseling is voluntary and that the nurse will also be available at the pharmacy to address concerns or questions whenever they arise outside of scheduled visits.
  Arms: Nurse-Navigator Enhanced PrEP Support

SUMMARY:
The investigators will conduct a cluster RCT in Kisumu, Kenya to determine the effect of nurse-navigators on PrEP initiation, persistence, and adherence among AGYW seeking contraception within a pharmacy-based PrEP delivery model. The study will randomize 20 retail pharmacies offering PrEP (10 pharmacies per randomization arm) and will enroll 1900 AGYW seeking contraception. All participants will be enrolled following purchase of a contraceptive method, offered PrEP (daily oral PrEP or the DPV-VR) and followed for 10 months. The study will quantify and compare PrEP initiation, persistence, and adherence at the pharmacy-level between randomization arms, in addition to several secondary and exploratory outcomes.

DETAILED DESCRIPTION:
In Aim 1, the investigators will conduct a cluster RCT in Kisumu, Kenya to determine the effect of nurse-navigators on PrEP initiation, persistence, and adherence among AGYW seeking contraception within a pharmacy-based PrEP delivery model. The study will randomize 20 retail pharmacies offering PrEP (10 pharmacies per randomization arm) and will enroll 1900 AGYW seeking contraception. All participants will be enrolled following purchase of a contraceptive method, offered PrEP (daily oral PrEP or the DPV-VR) and followed for 10 months. The study will quantify and compare PrEP initiation, persistence, and adherence at the pharmacy-level between randomization arms, in addition to several secondary and exploratory outcomes.

Pharmacy selection for cluster RCT (Aim 1): The investigators conducted a landscape analysis of all pharmacies in Kisumu, Kenya as part of the team's ongoing pharmacy-based PrEP delivery studies. In this analysis, the investigators gathered information on the types of customers who attend pharmacies, the types of services offered (e.g., HIV testing) and products purchased (e.g., contraceptive methods) at pharmacies, and availability of a separate private consultation room. The investigators will select 20 pharmacies based on whether they are willing to provide PrEP per national guidelines, have a separate consultation room that can be used for HIV testing and PrEP counseling, and provide the full range of contraceptives to AGYW clients (including EC, OCP, injectables, implants, and condoms).

Randomization (Aim 1): All the pharmacies will receive standard pharmacy-based PrEP delivery and be randomized to either receive (n=10 pharmacies) or not receive (n=10 pharmacies) a nurse-navigator to assist with PrEP delivery. To ensure balance between randomization arms in terms of key site characteristics, sites will be categorized on AGYW volume (i.e., monthly number of purchases made by AGYW clients) and distribution frequency of contraceptive methods purchased (based on pharmacy log data) and restricted randomization will be used for site (cluster) allocation to intervention and control arms. Specifically, all possible randomizations that evenly distribute sites on these specified factors (AGYW client volume and distribution of contraceptive methods) into 2 study arms will be generated, and one combination will be selected using a random number generator. Randomization and allocation will be performed by a biostatistician from the UW CFAR Biometrics Core, who has no knowledge of sites other than the variables included in the restricted randomization process, and the Study Statistician, who received an MPH in Biostatistics from UW, will supervise the randomization process. Once assigned, the randomization allocation will be unblinded. Since the randomization will occur at the pharmacy level, it is impossible to blind study team members or participants to the randomization assignments. However, procedures to minimize the influence of the unblinded nature of this study on outcomes will be implemented. Ongoing data monitoring will not include information about study endpoints disaggregated by site or study arm. Only the study statistician will review data on study endpoints by study arm or facility.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Seeking contraception (EC, OCP, injectables, implants, and condoms) from the retail pharmacy site
* Age between ≥14 and <25 years old
* Willingness to receive PrEP screening per national guidelines including HIV testing
* Not currently taking PrEP
* Able and willing to provide informed consent for participation

Exclusion Criteria:

* Male gender
* Not seeking contraception (EC, OCP, injectables, implants, and condoms) from the retail pharmacy site
* Age <14 and >24 years old
* Not willing to receive PrEP screening per national guidelines including HIV testing
* Currently taking PrEP
* Not able and/or willing to provide informed consent for participation

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1900 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
PrEP initiation | At enrollment
  Binary endpoint (Yes/No) based on self-reported use of daily oral PrEP pills or the DPV-VR at 1-month follow-up after acceptance at enrollment. Self-reported PrEP use will be considered initiation. If a participant declined PrEP at enrollment or reported not using PrEP after acceptance, the participant will be considered non-initiated
PrEP persistence | at 10 months
  Binary endpoint (Yes/No) based on self-reported persistent use of daily oral PrEP pills or the DPV-VR at 10-month follow-up after initiation at 1-month follow-up. Self-reported PrEP use will be considered persistence. If a participant declined PrEP at enrollment or reported not using PrEP after acceptance or discontinued PrEP before 10 months, the participant will be considered non-persistent
PrEP adherence | at 10 months
  Binary endpoint (Yes/No) based on hair samples from 10-month visits. Detectable TFV levels in hair >0.038 ng/mg or DPV levels >0.0248 n/mg will be considered adherent. If a participant stopped PrEP use or exited the study before 10 months (ie no hair sample collected), the participant will be considered non-adherent

SECONDARY OUTCOMES:
PrEP method selection | At enrollment
  Binary endpoint (Yes/No) of self-selection of DPV-VR compared to daily oral PrEP when offered at enrollment
Predictors of non-adherence | at 10 months
  Factors associated with poor adherence (outcomes of <90% adherent on PrEP or discontinuation) will include demographics, relationship/partner characteristics, psychosocial factors, socioeconomic status, low health/HIV literacy, fear of disclosure
STI incidence | at 10 months
  Frequency of STI (syphilis, gonorrhea, chlamydia) detection at follow-up visits will be compared between randomization arms

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Pintye, PhD, Principal Investigator — University of Washington
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya

REFERENCES:
- [Derived] Lagat HK, Pintye J, Harrington E, Houck S, Kwena Z, Lenn M, Mogaka F, Momanyi V, Mugambi M, Nyerere B, Odoyo J, Omollo V, Ortblad KF, Rota G, Sharma M, Bukusi EA. Enhancing HIV pre-exposure prophylaxis outcomes among Kenyan adolescent girls and young women with a novel pharmacy-based PrEP delivery platform: protocol for a cluster-randomized controlled trial. Trials. 2024 Jun 19;25(1):394. doi: 10.1186/s13063-024-08206-6. PMID 38890744